CLINICAL TRIAL: NCT01093898
Title: The Neuroeconomics of Behavioral Therapies for Adolescent Substance Abuse
Acronym: Imaging
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Catherine Stanger, Associate Professor, Dartmouth-Hitchcock Medical Center
Other Study IDs: 36824; 1R21DA029442-01 (NIH)
Record Dates: First submitted 2010-03-23; First posted 2010-03-26 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Adolescent Substance Use

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No intervention

SUMMARY:
This study will measure the brain activity of adolescent substance abusers while they make decisions about their preferences to receive smaller, immediate rewards versus larger delayed rewards. The investigators expect that patterns of brain activity while engaged in this decision making task will predict response to treatment among adolescent substance users. The investigators expect to use the results of this study to develop more effective treatments for adolescent substance abuse

DETAILED DESCRIPTION:
Little is known about the role of adolescent neurodevelopment in adolescent substance abuse treatment outcomes. The development and evaluation of adolescent substance abuse treatments rarely includes consideration of varying cognitive capacities and their neural representations as determinants of individual variation in treatment response. This proposed R21 project would address this gap by identifying associations among decision making, task-related neural processing, and treatment outcome among adolescents participating/have participated in two randomized clinical trials for adolescent substance abuse. Increasing our understanding of neural processes that underlie decision making in adolescent marijuana and alcohol users would inform the development of future intervention and prevention efforts.

This complementary project draws subjects from two studies investigating contingency-management (CM) based treatments "Behavioral Treatment of Adolescent Marijuana Abuse" (DA015186), and "Family Based Contingency Management for Adolescent Alcohol Abuse" (AA016917). Both trials compare a unique CM intervention that involves an abstinence-based reinforcement program to a standard, state of the art cognitive behavioral intervention. Analyses would be performed separately for the two samples, with hypotheses tested first using the Marijuana sample, and assessed for replication/specificity using the Alcohol sample. The proposed project would explore novel neurobiological predictors of response to CM interventions.

Adolescents recruited into the Marijuana Trial (n=69; 23 per treatment arm) and the Alcohol Trial (n=54; 27 per treatment arm) during the period of this R21 project would participate in a single neuroimaging session as soon after the intake session as possible, within 7 to 30 days. During the neuroimaging session, adolescents would make intertemporal choice decisions in a Delay Discounting task regarding gains of $100 and $1,000. Preliminary data from the Marijuana trial demonstrates significant association between performance on this behavioral delay discounting task and abstinence achieved during treatment over and above the significant effect of treatment condition. The investigators seek to understand the neural processes that underlie performance on this laboratory task, and the degree to which variation in these neural processes relates to and predicts adolescent substance abuse treatment outcomes. The conceptual framework for the proposed project is based on the neuroeconomics of addiction in general, and the competing neural systems hypothesis in particular (Bechara, 2005a; Bickel, et al., 2007; Daw, et al., 2005; Jentsch & Taylor, 1999). This behavioral choice hypothesis postulates a biased competition between an "impulsive" (or ''reflexive") neural system (including the striatum, amygdala, ventral pallidum, and related structures) and the "executive" (or "reflective") neural system (including the prefrontal cortex) in understanding patterns of suboptimal decision making among substance-dependent individuals. An overarching hypothesis is that differing responses to distinct treatment approaches (CM vs. CBT) are partially determined by the pattern of activation or functional connectivity within and across these competing neural systems. These project hypotheses would be tested by the following specific aims:

Primary Aims:

* Determine the degree to which performance on a laboratory delay discounting task correlates with activity in impulsive and/or executive neural systems.
* Determine the degree to which performance on a laboratory delay discounting task and neural processing predict adolescent substance abuse treatment outcome over and above the effects of treatment condition.

Secondary Aim:

* Explore interactions between response to CM and delay discounting-related neural processing.

In summary, this proposed exploratory/developmental project would importantly contribute to the understanding of the role of neural processing in adolescent substance-abuse treatment processes and outcome. Specifically, this study has the potential to reveal relations among decision making, neural processing, and treatment outcomes, including the role of patterns of neural activation on response to contingency management among adolescent substance abusers. Results will have implications for future research on adolescent neurodevelopment and adolescent substance abuse treatment. The potential to use neuroscience findings to better understand and improve treatment outcomes in substance-abusing adolescents will have strong public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 12 to 18 years old and have a parent/guardian who can participate.
* Youth must meet either of the following inclusion criteria:

  1. Report using marijuana during the previous 30 days or provide a marijuana-positive urine test, plus meet criteria for Cannabis Abuse or Dependence OR
  2. Meet Diagnostic Statistical Manual (DSM) criteria for Alcohol Abuse or dependence or have had one binge episode, specified by ≥5 drinks in one day, in the past 90 days and report alcohol use in the past 30 days.

Exclusion Criteria:

* Contraindications to MRI including ferromagnetic implants or claustrophobia
* Meeting DSM criteria for dependence on illicit drugs other than marijuana or alcohol (use/abuse of other drugs will not be excluded)
* Exhibit active psychosis, have severe medical or psychiatric illness limiting participation
* Are pregnant or breast-feeding.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents recruited into the Marijuana Trial and the Alcohol Trial during the period of the R21 project would participate in a single neuroimaging session as soon after the intake session as possible.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
delay discounting | Assessed at baseline
  laboratory task assessing preference for immediate rewards

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Stanger, Ph.D., Principal Investigator — Dartmouth College
Locations (1):
- Geisel School of Medicine at Dartmouth, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stanger C, Elton A, Ryan SR, James GA, Budney AJ, Kilts CD. Neuroeconomics and adolescent substance abuse: individual differences in neural networks and delay discounting. J Am Acad Child Adolesc Psychiatry. 2013 Jul;52(7):747-755.e6. doi: 10.1016/j.jaac.2013.04.013. Epub 2013 Jun 5. PMID 23800488